CLINICAL TRIAL: NCT00949611
Title: Wiser Choices In Osteoporosis Choice II
Brief Title: Wiser Choices in Osteoporosis Choice II: A Decision Aid for Patients and Clinicians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Foundation for Informed Medical Decision Making (Other); Olmsted Medical Center (Other)
Responsible Party: Principal Investigator, Victor Montori, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 08-006070
Record Dates: First submitted 2009-07-28; First posted 2009-07-30 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Osteoporosis; Osteopenia; Fragility Fractures
Keywords: Decision Aid; Shared Decision Making; Shared Medical Decision Making
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic | interventions — Decision Support Techniques

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- FRAX + Decision Aid (Experimental)
  Interventions: Behavioral: FRAX + Decision Aid
- Usual care (No Intervention)
- FRAX estimated fracture risk (Experimental)
  Interventions: Behavioral: FRAX estimated fracture risk

INTERVENTIONS:
Behavioral: FRAX + Decision Aid — Clinicians will present patient's with their individualized risk of osteoporotic fracture in 10 years, based on the FRAX risk calculator, as well as sharing a decision aid with them, which shows their risk of fracture, risk reduction on medications, as well as the downsides of the medications.
  Other Names: Decision Support
  Arms: FRAX + Decision Aid
Behavioral: FRAX estimated fracture risk — The clinician is provided with the patient's estimated risk of fracture as computed by the FRAX
  Other Names: Risk estimate
  Arms: FRAX estimated fracture risk

SUMMARY:
Emphasis in treating osteoporosis has been on T-scores rather than overall fracture risk. Fracture Risk Assessment Tool (FRAX) supports a risk sensitive approach to osteoporosis treatment by providing an absolute fracture risk. FRAX combined with a decision aid may promote a shared decision making approach with patients, allowing the clinician and patient to weigh potential fracture risk (without treatment), versus risk reduction with medication (including side effects and costs). OSTEOPOROSIS CHOICE II will test the effectiveness of:

* FRAX
* FRAX + decision aid
* Usual care (no decision aid and no FRAX given to clinician)

ELIGIBILITY:
Inclusion Criteria:

* Peri and Postmenopausal Caucasian, Black, Hispanic and Asian women, aged 50-90
* Bone mineral density (BMD) T-Score < 1.0
* Have appointment with clinician to discuss test results and treatment options
* Patients with FRAX <20% risk who have taken a bisphosphonate for < 5 years.

Exclusion Criteria:

* Unable to speak or read English

Ages: 50 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2009-05; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Medication start/stop, knowledge, and patient involvement. | Baseline and at 6 months

SECONDARY OUTCOMES:
Decisional quality. | Baseline and at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Victor M. Montori, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] LeBlanc A, Wang AT, Wyatt K, Branda ME, Shah ND, Van Houten H, Pencille L, Wermers R, Montori VM. Encounter Decision Aid vs. Clinical Decision Support or Usual Care to Support Patient-Centered Treatment Decisions in Osteoporosis: The Osteoporosis Choice Randomized Trial II. PLoS One. 2015 May 26;10(5):e0128063. doi: 10.1371/journal.pone.0128063. eCollection 2015. PMID 26010755
- [Derived] Wyatt KD, Branda ME, Inselman JW, Ting HH, Hess EP, Montori VM, LeBlanc A. Genders of patients and clinicians and their effect on shared decision making: a participant-level meta-analysis. BMC Med Inform Decis Mak. 2014 Sep 2;14:81. doi: 10.1186/1472-6947-14-81. PMID 25179289